CLINICAL TRIAL: NCT02920918
Title: A Randomized Active-Control Double-Blinded Study to Evaluate the Treatment of Diabetes in Patients With Systolic Heart Failure
Brief Title: Treatment of Diabetes in Patients With Systolic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20007043; 28431754DIATBD (Other Grant/Funding Number: Janssen Scientific Affairs)
Record Dates: First submitted 2016-09-22; First posted 2016-09-30 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure, Systolic; Diabetes Mellitus, Type 2
Keywords: Systolic Heart Failure; Canagliflozin; Sitagliptin Phosphate; Type 2 Diabetes; SGLT2 inhibitor; DPPIV inhibitor
MeSH Terms: conditions — Heart Failure, Systolic; Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canagliflozin (Active Comparator): Canagliflozin will be administered orally in pill form at 100 mg, daily for 12 weeks.
  Interventions: Drug: Canagliflozin
- Sitagliptin (Active Comparator): Sitagliptin will be administered orally in pill form at 100 mg, daily for 12 weeks.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Canagliflozin
  Other Names: Invokana
  Arms: Canagliflozin
Drug: Sitagliptin
  Other Names: Januvia
  Arms: Sitagliptin

SUMMARY:
Investigator Initiated Study to study the effects of Canagliflozin 100 milligrams (mg) vs Sitagliptin 100 mg on parameters of aerobic exercise capacity (peak oxygen consumption [VO2]) and ventilator efficiency (minute ventilation [VE]/carbon dioxide production [VCO2] slope) at cardiopulmonary exercise test (CPET) after 12 weeks of active treatment (primary endpoints). Blood pressure (BP), body water content, body composition, cardiac function, and diet will be also measured (secondary endpoints).

DETAILED DESCRIPTION:
Investigator Initiated Study: Randomized, double-blinded, active-control clinical trial to determine the safety and efficacy of Canagliflozin and Sitagliptin in patients with type 2 diabetes and systolic heart failure (HF).

The investigators propose to study the effects of Canagliflozin 100 mg vs Sitagliptin 100 mg (both administered once daily for 12 weeks) on parameters of aerobic exercise capacity and ventilator efficiency by CPET after 12 weeks of active treatment. BP, body water content (Bioelectrical Impedance Analysis [BIA]), body composition (Dual-energy X-ray absorptiometry [DEXA]), cardiac function, diet and biomarkers will be also measured. Subjects with evidence of left ventricular hypertrophy will undergo cardiac magnetic resonance (CMR) imaging.

ELIGIBILITY:
Major Inclusion Criteria:

* Symptomatic stable heart failure (New York Heart Association (NYHA) functional classification II-III) with reduced left ventricular ejection fraction (LVEF) ≤40%
* Peak exercise limited by shortness of breath and associated with a respiratory exchange ratio (RER) >1.00 (reflecting maximal aerobic effort);
* Poorly controlled Type 2 Diabetes Mellitus (T2DM)(HbA1c levels between 7.0% and 10.0% if on a treatment regimen including insulin, or between 6.5% and 10.0% if not on an insulin regimen);
* Eighteen years of age or older.

Major Exclusion Criteria:

* Type I diabetes;
* Open label treatment with Sodium-GLucose coTransporter (SGLT)-2 inhibitors (within the past 3 months);
* Current treatment with thiazolidinedione (within the past 3 months);
* Chronic Renal Disease defined as Glomerular Filtration Rate (GFR) <50 ml•min-1/1.73m2 according to local laboratory
* Pregnancy or of child-bearing potential or lactating;
* Active or recent (within 2 weeks) genital/urinary infection;
* Concomitant conditions or treatment which would affect completion or interpretation of the study (i.e, physical inability to walk or run on a treadmill
* Inability to give informed consent.

Exclusion criteria specific to the cardiac magnetic resonance (CMR) substudy.

* Estimated GFR <60 ml•min-1/1.73m2
* Implantable cardioverter defibrillator, pacemaker or other implantable metal device not compatible with CMR scanning;
* Severe claustrophobia, inability to lay flat for up to 60 minutes, or other contraindication to CMR scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to present the data promptly upon analysis as an abstract to a national meeting and/or a manuscript.
Supporting Information: CSR
Time Frame: Data were presented as late breaking clinical trial at the Heart Failure Society of America (HFSA) 2019 in Philadelphia as poster presentation.
Access Criteria: Data in the form of poster were made available from HFSA.
URL: https://www.eventscribe.com/2019/HFSA/PosterTitles.asp?pfp=PosterTitles

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin: Canagliflozin will be administered orally in pill form at 100 mg, daily for 12 weeks.
  Canagliflozin
- Sitagliptin: Sitagliptin will be administered orally in pill form at 100 mg, daily for 12 weeks.
  Sitagliptin
Period: Overall Study
Arm/Group | Canagliflozin | Sitagliptin
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canagliflozin | Sitagliptin | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 19 | 34
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.1) | 54.3 (8.8) | 56.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36
Peak Oxygen Consumption [Mean (Standard Deviation); unit: mL/kg/min] — Peak oxygen consumption (VO2) measured with maximal cardiopulmonary exercise test.
  mL/kg/min | 16.2 (3.4) | 15.3 (3.5) | 15.7 (3.4)
Ventilator Efficiency [Mean (Standard Deviation); unit: Unitless] — Minute ventilation (VE) relative to CO2 production (VCO2) slope measured by cardiopulmonary exercise test
  Unitless | 34.1 (6.1) | 32.6 (7.2) | 33.3 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Aerobic Exercise Capacity at 12 Weeks
Description: Peak oxygen consumption (VO2) measured by maximal cardiopulmonary exercise test
Time Frame: baseline and 12 weeks
Population: Unadjusted p values were reported throughout, with statistical significance set at the 2-tailed 0.05 level. Only cases with available data used to compute the primary endpoint will be included in the analyses (16 subjects for canagliflozin group and 18 subjects for sitagliptin group).
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Canagliflozin | Sitagliptin
Number analyzed (Participants) | 16 | 18
mL/kg/min | 0.67 (2.10) | -0.53 (1.75)
Statistical Analysis 1: Comparison: Canagliflozin vs Sitagliptin; We expected a baseline peak oxygen consumption (VO2) of 14.5 mL/kg/min. A sample size of 40 patients per group (total of 80 patients) provided sufficient power to detect a mean difference in the interval change in peak VO2 of 1.50±1.76 mL/kg/min (primary endpoint) expected with Canagliflozin compared to Sitagliptin, which we predict to have no significant effect on peak VO2 (0±1.76 mL/kg/min); Test type: Superiority; p = 0.083, ANOVA

2. Primary Outcome: Change From Baseline Ventilatory Efficiency at 12 Weeks
Description: Minute ventilation (VE) relative to CO2 production (VCO2) slope measured by cardiopulmonary exercise test
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Canagliflozin | Sitagliptin
Number analyzed (Participants) | 16 | 18
Unitless | -0.3 (4.1) | -0.3 (5.1)
Statistical Analysis 1: Comparison: Canagliflozin vs Sitagliptin; Test type: Superiority; p = 0.51, ANOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An event that is considered by the investigator(s) to be expected and related to the natural history of the disease is not considered an AE.
Arm/Group | Canagliflozin | Sitagliptin
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/17 | 1/19
Other Adverse Events (participants affected / at risk) | 7/17 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canagliflozin (N=17) | Sitagliptin (N=19)
Influenza B (Infections and infestations) | 0 (0) | 1 (1)
Occlusion superficial femoral artery (Vascular disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness and acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canagliflozin (N=17) | Sitagliptin (N=19)
Genital infection (Infections and infestations) | 1 (1) | 1 (1)
Hypotensive event (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmic events (Cardiac disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02920918/Prot_SAP_ICF_000.pdf